| A Single-Center Trial to Evaluate the Efficacy and Tolerability of the SkinPen | |
|---|---|
| SPONSOR STUDY NUMBER: | Bellmed002 |
| SPONSOR: | Bellus Medical |
| SPONSOR'S REPRESENTATIVE: | |
| TESTING AND ADMINISTRATIVE FACILITY: | |
| INVESTIGATOR: | |
| SUB-INVESTIGATOR/STUDY PHYSICIAN: | |
| SUB-INVESTIGATOR: | |
| DATE: | |

# A Single-Center Trial to Evaluate the Efficacy and Tolorability of the Skin Day SIGNATURE PAGE

Investigator

Sub-Investigator/Study Physician

Sub-Investigator .

Sub-Investigator

Sponsor Representative Bellus Medical

Date

Version #2.0

# A Single-Center Trial to Evaluate the Efficacy and Tolerability of the SkinPen SIGNATURE PAGE

| Date | | |
|---|---|---|
| Date | | Date |
| Date | Part Control of the C | |
| | | Date |
| Date | | Date |
| Date | | |
| | | Date |

Study Number: Bellmed002

Version #2.0

#### **TABLE OF CONTENTS**

| | Page |
|-----|------|
| 100 | |
| _ | |
| _ | |
| _ | |
| Ξ, | |
| 7 | |
| _ | |

CONFIDENTIAL Bellus Medical

Study Number: Bellmed002 Version #2.0

| 10. | ADVERSE EVENTS | 20 |
|-----------|-------------------------------------|----|
| 10 | 0.1. Definition of an Adverse Event | 20 |
| :<br>: | | |
| 15.<br>15 | BIOSTATISTICS AND DATA MANAGEMENT | |

| RP |
|----|

| This single-center, clinical trial is being conducted over the course of 90 days post-treatment visits in order to assess the efficacy and tolerability of the Sponsor's SkinPen device when used by men and women with |
|---|
| 3. HYPOTHESIS |
| The Sponsor's test materials will produce a statistically significant improvement in appearance over the course of 90 days of use (4 monthly treatments), |
| 4. STUDY ENDPOINTS |
| 4.1. Primary Endpoints |
| Assessment of wrinkles severity using a Lemperle Wrinkle Assessment Scale |
| 3-month post-treatment. |
| Monitoring of adverse events throughout the course of the study. |
| Subjects global aesthetic improvement assessment at |
| Patient Satisfaction Questionnaire |
| <ul> <li>Measurements to assess skin thickness, skin density and firmness using the OCT, ultrasound<br/>and BTC 2000 respectively.</li> </ul> |
| 5. TEST MATERIAL INFORMATION |
| 5.2 Characterization and Stability |

### 5.2. Characterization and Stability

The Sponsor assumes responsibility for chemical characterization and stability of the study device(s).

# 5.3. Study Device Description(s)

| | 100 | | 54 87 |
|---|---|---|---|
| IL. | DOLOTO DOO, HOMEO, FORMING OPEN | 0011101000 | or, mod o, oo Lo to doon |
| D | Pollus Modical | | 15. 22.23 |

Bellus Medical Study Number: Bellmed002

Version #2.0



#### **5.4. Method of Treatment Assignment**

Subjects will be numbered sequentially in the order in which they qualify for entry into the study. Prior to the start of the study, all subjects will receive treatment with the device as outlined in the instructions.

#### 5.5. Study Device Accountability

Upon receipt of the clinical supplies at the site, designated study personnel will conduct a complete inventory of all study devices and assume responsibility for their storage and dispensation.

All supplies sent to the study site will be accounted for and in no case will be used

Used and unused devices will be returned to the Sponsor. Documentation will be provided for any devices not returned by subjects in the study file.

#### 5.6. Storage of Study Devices

The Investigator will agree to keep all study devices in a safe and secure area with restricted access in accordance with applicable regulatory requirement(s).

#### 5.7. Treatment Compliance

Any suspected non-compliance will be addressed by the Investigator or designee. The Investigator will make a determination if a subject's non-compliance will have an effect the outcome of the study and if the subject should be dropped from the study and/or data should be excluded from statistical analyses.

#### 6. SUBJECT ENROLLMENT AND INSTRUCTIONS

#### 6.1. Number of Subjects

At least 33 subjects meeting the eligibility requirements are expected to complete participation in the clinical trial.

| | 6.1.1. <u>Determination of Sample Size</u> The sample size determination of this study |
|---|---|
| 6.2 | Informed Consent Form |
| | An IRB-approved informed consent form (ICF), |

| An IRB-approved informed consent form (ICF), |
|---|
| will be given to each candidate subject before participation in ar |
| study procedures. The candidate subject will be given as much time as needed to read the ICF ar |
| will have the opportunity to have any study related questions answered to their satisfaction prior |
| signing the ICF. |

Bellus Medical Study Number: Bellmed002 Version #2.0 CONFIDENTIAL

#### 6.3. Subject Identification



#### 6.4. Eligibility Criteria

Individuals will be admitted to the study at the discretion of the Investigator or designee, based on medical history and findings of the pre-study interview and examination. Individuals will be screened for the eligibility criteria listed below prior to study enrollment.

#### 6.4.1. Inclusion Criteria




Study Number: Bellmed002 Version #2.0





#### 6.5. Subject Instructions

Subjects will be provided with the following instructions to follow during the study:



To keep skincare product consistency, Subjects will be offered

Sunscreen is recommended to be applied each morning and prior to any sun exposure.

#### 6.5.3. Subject Instructions for Study Visits

 Remove all makeup at least 30 minutes prior to each scheduled clinic visit using the provided facewash.

#### 6.5.4. General Study Instructions

 Avoid extended periods of sun exposure and all use of tanning beds for the duration of the study. Extra care should be taken to wear protective clothing, including sunglasses, and avoid sun exposure from 10 AM to 4 PM.



#### 7. STUDY DESIGN

#### 7.1. Description

This is a study to evaluate the efficacy of the microneedling device in improving

Overall assessment of clinical outcome and safety will be based on clinic visits and evaluation of pre- and post- procedural photos. These photos will be and subjects will be adequately informed of such. In conjunction with standard and close-up photography,

high-resolution ultrasonography, optical coherence tomography, transepidermal water loss measurements, and/or


Study Number: Bellmed002 Version #2.0



#### 7.2. Outline of Procedures



#### 7.3.



#### 8. CONDUCT OF STUDY

#### 8.1. Pre-Study Procedures

- Prior to the start of the study, prospective subjects will be screened for eligibility requirements by telephone.
- 2. Prospective subjects will be informed of the pre-study washout phase pre-visit procedures as described in sections 5.5.1 and 5.5.3.

3. Prospective subjects will be assigned an appointment time for visiting the clinic.

| 8.2. Baseline: | Visit 1 | (-14 to | 0 day[s]) |
|----------------|---------|---------|-----------|
|----------------|---------|---------|-----------|

- Candidate subjects will be given an IRB-approved informed consent form (ICF)
- 2. Candidate subjects will complete an eligibility and health questionnaire.
- 3. Candidate subjects that sign the initial paperwork will be assigned a screening number.
- Candidate subjects will be screened by the Investigator or designee for qualification criteria.
- Candidate subjects that pass the initial screening will be graded for wrinkle severity and as described in section 8.1.
- Those that pass eligibility requirements and are female will perform a pregnancy test (if necessary); if the test is negative or the candidate subject is male, the subject will be enrolled into the study and assigned a subject number.

| 8.3. In | terim Visits: Visits 2-5 |
|---|---|
| | A clinician will record concomitant medications and will ask subjects if they have experienced any changes in their health since the previous visit. |
| 3. | After acclimation, subjects will participate in TEWL Measurements, OCT images, high frequency ultrasounds images, BTC images and imaging procedures as described in section |
| 5. | Trained aestheticians will treat |

8.4. Post-Treatment Visit: Visit 6

diaries will be distributed at Visit

A clinician will record concomitant medications and will ask subjects if they have experienced any changes in their health since the previous visit.

6. Subjects will be provided with supporting materials, usage instructions and a daily diary. New

| 2. | Supporting products and daily diary distributed at Visit will be reviewed for compliance. |
|---|---|
| 3. | After a 15 minute acclimation to ambient temperature and humidity conditions, subjects will participate in the following procedures: • Imaging procedures as described in section |
| | <ul> <li>Assessment of Wrinkle</li> <li>Clinician's global aesthetic improvement assessment as described in section</li> <li>Subject's self-assessment on improvement as described in section</li> <li>Patient Satisfaction Questionnaire as described in section</li> <li>TEWL measurement, OCT images, high frequency ultrasound images and BTC 2000 measurement.</li> </ul> |
| 8.5. Po | st-Treatment Visit: Visit 7 |
| 1. | A clinician will record concomitant medications and will ask subjects if they have experienced any changes in their health since the previous visit. |
| 2. | Subjects will participate in pregnancy screening procedures. |
| 3. | After a 15 minute acclimation to ambient temperature and humidity conditions, subjects will participate in the following procedures: • Imaging procedures as described in section |
| | <ul> <li>Assessment wrinkle</li> <li>Clinician's global aesthetic improvement assessment as described in section</li> <li>Subject's global aesthetic improvement as described in section 8.2.2</li> <li>Patient Satisfaction Questionnaire as described in section 8.6.</li> <li>TEWL measurement, OCT images, high frequency ultrasound images and BTC 2000 measurement.</li> </ul> |
| | <u></u> |

#### ASSESSMENTS

Note that the order of the assessment listed below may be altered from the order indicated in the study visits in order to help study flow, or at the recommendations of the Sponsor or Investigator. Any change in the order of procedures will not compromise study data.


Study Number: Bellmed002

Version #2.0

9.1. Assessment Wrinkling

Assessment of wrinkling will be performed at will be performed at will be assessed according to the following definitions:

Class 0: No Wrinkles

Class 1: Just perceptible wrinkle

Class 2: Shallow wrinkles

Class 3: Moderately deep wrinkle

Class 4: Deep wrinkle, well-defined edges Class 5: Very deep wrinkle, redundant fold



Study Number: Bellmed002 Version #2.0



#### 9.2. Global Aesthetic Improvement Assessment

#### 8.2.1 Clinician's Global Aesthetic Improvement Scale (CGAIS)

| Rating | Description |
|---|---|
| 1 | Very Much Improved: Optimal cosmetic result in this subject. |
| 2 | Much Improved: Marked improvement in appearance from the initial condition but not completely optimal for this subject. |
| 3 | <b>Improved:</b> Obvious improvement in appearance from initial condition, but a retreatment is indicated. |
| 4 | No Change: The appearance is essentially the same as the original condition. |
| 5 | Worse: The appearance is worse than the original condition. |

# 8.2.2 Subject Global Aesthetic Improvement Scale (SGAIS)

| Rating | Description |
|---|---|
| 1 | Very Much Improved: Optimal cosmetic result. |
| 2 | Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal. |

STU062018-069, Kenkel, FormA3-Sponsor Protocol, Mod\_6, 09-25-19 docx

© Bellus Medical


Study Number: Bellmed002

Version #2.0

| 3 | Improved: Obvious improvement in appearance from initial condition. |
|---|---|
| 4 | No Change: The appearance is essentially the same as the original condition. |
| 5 | Worse: The appearance is worse than the original condition. |

## 9.3. Imaging Procedures

| Prior to photography procedures, clinic personnel will ensure that subjects neck as described in the study procedures. Subjects will remove any jewelry from the area(s) to be photographed and equilibrate for at least 15 minutes to ambient conditions within the clinic before any photographs are taken. |
|---|
| Subjects will be provided with a black matte t-shirt or a black or gray matte cloth will be draped over the subjects' clothing. |
| 9.3.2. NIKON D7100 Standard, close-up and cross-polarized photography of process and the control of pr |

#### 9.4. Noninvasive Procedures

#### 9.6. Patient Satisfaction Questionnaires

Subjects will complete a Sponsor-provided self-assessment questionnaire

#### 10. ADVERSE EVENTS

#### 10.1. Definition of an Adverse Event

An adverse event (AE) is any untoward medical occurrence in a clinical investigation where a subject is administered a pharmaceutical product/biologic (at any dose), OTC, cosmetic product or medical device and which does not necessarily require a causal relationship with a test article.

#### 10.2. Assessment of Severity and Relationship

The Investigator or medical staff will evaluate all AEs as to their severity and relation to the test article.

The severity of an AE will be graded as follows:

Mild: Awareness of a sign or symptom but easily tolerated

Moderate: Discomfort sufficient to cause interference with usual activity or to affect clinical

status

Severe: Incapacitating with inability to do usual activity or to significantly affect clinical

status



#### 10.3. Definition of a Serious Adverse Event

A serious adverse event (SAE) is any experience or reaction occurring at any dose that results in any of the following outcomes:

- death,
- is life threatening.
- inpatient hospitalization or prolongation of hospitalization,
- a persistent or significant disability/incapacity, or
- a congenital anomaly/birth defect.

Bellus Medical Study Number: Bellmed002 Version #2.0

| 10.4. Procedures for Reporting Adverse Events |
|---|
| At each visit, the Investigator or designee will question the subject about adverse events using ar<br>open question and taking care not to influence the subject's answer (e.g. "Have you noticed any<br>change in your health since the last visit?"). |
| The Sponsor will be notified of all AEs within 5 business days. Photographs will be taken to documen any AEs if possible. |
| 10.5. Procedures for Reporting Serious Adverse Events |
| Any SAE that occurs during the study whether related to the treatment or not, expected or not, will be reported to the Sponsor Representative immediately (within 24 hours of being reported to the Investigator) |
| 10.6. Procedures for Reporting Pregnancies |
| All pregnancies occurring during clinical studies must be reported to the Sponsor by the Investigato within 24 hours of observation or notification of the occurrence. |
| 10.7. Medical Treatment for Adverse Events and Serious Adverse Events |

12. ADVERSE WEATHER PROVISION

#### 13. PROTOCOL MODIFICATIONS

Protocol amendments will be written to record any changes or formal clarification to the procedures outlined in the protocol. Any violations to the protocol that might significantly affect the completeness, accuracy and/or reliability of the study data or might affect the subjects' rights, safety or well-being will be documented as protocol deviations.

| additionated as protocol astractions. |
|---|
| All protocol amendments will be forwarded to the IRB for review and approval prior to implementation even if it is determined the safety of the subjects will not be affected. |
| 14. ETHICAL AND REGULATORY PROCEDURES |
| 14.1. Research Standards/Good Clinical Practice |
| The conduct of this study will follow all applicable guidelines for the protection of human subjects for research as outlined in 21 CFR 50, in accordance with the accepted standards for Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and the standard practices of Un Southwestern |
| 14.2. Quality Control and Quality Assurance |
| The Investigator will permit trial-related monitoring, audits, IRB review, and regulatory inspection(s) by providing direct access to source data/documents. |
| 14.3. Institutional Review Board |
| This study (protocol, ICF and all addenda) will be reviewed and approved by an Institutional Review Board (IRB). The study will not be activated, subjects will not be consented or receive any study devices or participate in any study procedures until such time as the IRB has approved the protocol and the ICF. |
| 15. BIOSTATISTICS AND DATA MANAGEMENT |
| 15.1. Statistical Analysis Population |
| The per-protocol (PP) population will be the primary population for all statistical analyses. |
| The per protests (11) population will be the primary population for all stational analysis. |

# 15.2. Statistical Analysis Plan

| This initial study will include descriptive statistics and change from baseline analysis. | |
|---|---|
| A descriptive statistical summary severity using the Lemperle Wrink | will be provided for all clinical assessments (including wrinkle |
| Aquaflux, Vivosight, BTC 2000 m summary includes the number of company includes the number of | subjects global aesthetic improvement (SGAIS), |
| estimated at post-baseline time po | ne (defined as post-baseline value minus baseline value) will be<br>pints for applicable parameters. The null hypothesis, that the mean<br>be tested using methods described in the Statistical Analysis Plan |
| The following will be calculated as baseline time point(s): | nd reported for each evaluation parameter at the applicable post- |
| | from(visit mean score – baseline mean score) x 100 |
| baseline = | baseline mean score |
| Percent of subjects | (number of subjects improved/worsened from baseline) x 100 |
| improved/worsened = | total number of subjects |



All statistical tests will be 2-sided at significance level alpha=0.05. P-values will be reported to 3 decimal places (0.000). No multiple testing corrections will be considered in the study. Statistical analyses are performed using SAS software version 9.4 or later series (SAS Statistical Institute).



#### 16. CLINICAL STUDY REPORT

A clinical study report will be drafted using template and incorporating any documented Sponsor preferences on file. The draft report will be submitted to the Sponsor for approval prior to finalization, and revisions may be made at the Sponsor's request.



Bellus Medical
Study Number: Bellmed002

Version #2.0

#### 17. MAINTENANCE OF RECORDS

| Original records (including the study protocol, clinical grading records, medical histories, informed cons forms, screening/enrollment logs, and any other case report forms used in the study) and a copy of final study report will be retained on file gradient to a minimum or a minimum of the archiving time has expired, the study information will either be destroyed or sent to | the |
|---|---|
| Sponsor | |
| | 1 |
| | _ |
| | - |
| | i |
| | _ |

CONFIDENTIAL